CLINICAL TRIAL: NCT04048772
Title: Creating Affiliations, Learning, and Mindfulness for In Vitro Fertilization Patients
Brief Title: CALM IVF (Creating Affiliations, Learning, and Mindfulness for In Vitro Fertilization Patients)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rachel Whynott (Other)
Responsible Party: Sponsor-Investigator, Rachel Whynott, Fellow Physician, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201906788
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life; IVF; Patient Satisfaction; Patient Engagement; Patient Empowerment
Keywords: Relaxation; Education; Support; Group; Knowledge; Therapy; In vitro fertilization; Stress; Relationships; IVF
MeSH Terms: conditions — Patient Satisfaction; Patient Participation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standard of care in vitro fertilization patients randomized to the psychoeducational group intervention.
  Interventions: Behavioral: CALM IVF
- Control (Other): Standard of care in vitro fertilization patients at our institution.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: CALM IVF — The intervention will be three 1-1.5 hour interactive sessions that are scheduled throughout the participant's first in vitro fertilization cycle. These sessions will provide additional time for discussion about treatment with providers, learning opportunities on topics of interest to fertility patients, and stress reduction techniques.
  Arms: Intervention
Other: Standard of Care — Patients will receive the standard of care IVF treatment at the University of Iowa.
  Arms: Control

SUMMARY:
The investigators have designed a psychoeducational group curriculum specifically for new in vitro fertilization (IVF) patients (both male and female) to improve their treatment knowledge, to allow them to engage more in their care, to offer a support network, to improve satisfaction, and to provide them with tools to help reduce their stress and anxiety while undergoing the IVF process. The investigators plan to have four to eight infertility patients and their partners participate in a group at a time, for which they will attend three 1-1.5 hour interactive sessions that are scheduled throughout their first IVF cycle. These sessions will provide additional time for discussion about treatment with providers, learning opportunities on topics of interest to fertility patients, and stress reduction techniques. They will do several surveys before and after the intervention for comparison, including assessment of quality of life, depression, anxiety, resilience, and a knowledge assessment. The investigators will also track the patients to see if they pursue additional treatment in the instance of a negative pregnancy test compared to patients undergoing the standard treatment. The investigators plan to recruit a control group that receives the standard of care treatment here at the University of Iowa.

DETAILED DESCRIPTION:
Patients and their partners will be randomized in a 2:1 fashion to two different treatment arms: A) standard of care in vitro fertilization (IVF) at the investigational institution as well as participating in an additional psychoeducational group or B) standard of care IVF at the investigational institution. The intervention group will consist of three additional evening visits for 1-1.5 hours per session. The sessions will include an interactive educational component addressing usual questions and concerns of IVF patients, such as reviewing common IVF myths, and also more information regarding treatment and technologies. Each session will also include teaching of coping strategies (such as awaiting the pregnancy test, how to cope with insensitive remarks from friends and family) as well as relaxation exercises, such as progressive muscle relaxation and deep breathing.

The patients will be consented at their new IVF visit and will take their initial assessments (FertiQoL, GAD-7, PHQ-9, the Connor-Davidson Resilience Scale, and a knowledge assessment) within 24 hours of the new visit. The patients will be assigned into groups based on when they are going through their IVF stimulations, so they will have similar experiences at similar times. Patients will take their final assessments on the third day after egg retrieval, regardless of group assignment.

ELIGIBILITY:
Inclusion Criteria:

* All patients starting their first in vitro fertilization cycle at the University of Iowa Hospitals and Clinics

Exclusion Criteria:

* Patients who have already undergone in vitro fertilization treatment at any institution
* Non-English speakers
* Fertility preservation patients
* Patients using donor oocytes, embryos, or sperm
* Patients taking psychotropic medications for depression or anxiety that have had a dosing adjustment within 3 months of study enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in female fertility patient quality of life score during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  FertiQoL International (Fertility Quality of Life Questionnaire 2008), scored scale from 0-100, with higher values indicating a higher quality of life and low scores indicating a lower quality of life.

SECONDARY OUTCOMES:
Change in female GAD-7 score during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Generalized Anxiety Disorder 7-item scale, with higher scores indicating higher likelihood of an anxiety disorder and lower scores indicating less likelihood of an anxiety disorder.
Change in female PHQ-9 score during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Patient Health Questionnaire, with higher score indicating increased likelihood of a depressive disorder and lower scores indicating less likelihood of a depressive disorder.
Change in female Connor-Davidson Resilience Scale during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Connor-Davidson Resilience Scale, with higher scores indicating greater resilience, and lower scores indicating lower resilience
Change in female knowledge assessment during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Assessment of knowledge regarding IVF treatment, with higher scores indicating a greater knowledge of IVF treatment, and lower scores indicating less knowledge regarding IVF treatment
Likelihood of continued IVF treatment in the instance of a negative pregnancy test | Three months after embryo transfer
  Patients who are not pregnant after embryo transfer will be followed for three months to assess likelihood to return for additional treatment after negative embryo transfer outcome.
Change in male fertility patient quality of life score during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  FertiQoL International (Fertility Quality of Life Questionnaire 2008), scored scale from 0-100, with higher values indicating a higher quality of life and low scores indicating a lower quality of life.
Change in male GAD-7 score during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Generalized Anxiety Disorder 7-item scale, with higher scores indicating higher likelihood of an anxiety disorder and lower scores indicating less likelihood of an anxiety disorder.
Change in male PHQ-9 score during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Patient Health Questionnaire, with higher score indicating increased likelihood of a depressive disorder and lower scores indicating less likelihood of a depressive disorder.
Change in male Connor-Davidson Resilience Scale during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Connor-Davidson Resilience Scale, with higher scores indicating greater resilience, and lower scores indicating lower resilience
Change in male knowledge assessment during IVF treatment cycle | From enrollment to 2-4 days after oocyte retrieval
  Assessment of knowledge regarding IVF treatment, with higher scores indicating a greater knowledge of IVF treatment, and lower scores indicating less knowledge regarding IVF treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Whynott, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Whynott RM, Summers KM, Mejia RB, Segre LS, Ryan G, Pawlak SA. Creating affiliations, learning, and mindfulness for in vitro fertilization patients (CALM IVF): a clinical trial. F S Rep. 2023 Jan 7;4(1):61-71. doi: 10.1016/j.xfre.2023.01.002. eCollection 2023 Mar. PMID 36959953